CLINICAL TRIAL: NCT00376311
Title: Phase IIa Study of the Effects of a New Oral Formulation of Salmon Calcitonin in Human Osteoarthritis
Brief Title: Effects of Oral Salmon Calcitonin in Human Osteoarthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Daniel H Manicourt
Record Dates: First submitted 2005-12-30; First posted 2006-09-14 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2002-06

CONDITIONS: Osteoarthritis
Keywords: Lequesne's algo-functional score; Biomarkers of joint metabolism
MeSH Terms: conditions — Osteoarthritis | interventions — salmon calcitonin

INTERVENTIONS:
Drug: oral salmon calcitonin

SUMMARY:
To assess the safety, tolerability and clinical efficacy of oral salmon calcitonin in patients suffering from osteoarthritis

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a difficult condition to manage and, thus far, we have no simple, effective interventions for this common cause of pain and disability.

Because parenteral salmon calcitonin (sCT) has positive effects in canine experimental OA, this phase IIa, randomized,placebo-controlled, double-blind trial evaluates the safety, tolerance and clinical efficacy of an oral formulation of sCT in patients with OA.

Patients receive a tablet containing either a placebo, 0.5 mg sCT or 1 mg sCT that they have to take every day in the morning 15 minutes before breakfast for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* radiographic OA according to the criteria of the American College of Rheumatology;
* morning joint stiffness between 15 and 30 minutes;
* pain on weight bearing and motion reported greater than 40 mm on a 0-100 mm visual analogue scale;
* normal liver and kidney function tests;
* serum CRP levels < 10 mg/l

Exclusion Criteria:

* previous or ongoing treatment with anti-resorptive drugs such as bisphosphonates, estrogen or raloxifene
* crystal deposition diseases
* known hereditary or congenital defects
* clinically significant hepatic, renal, cardiovascular, psychiatric, endocrine and/or hematological diseases
* intra-articular injections of either corticosteroids (previous 3 months) or hyaluronan (previous 6 months)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2002-09; Study Completion 2004-05

PRIMARY OUTCOMES:
Lequesne's algofunctional index
Biomarkers of joint metabolism

SECONDARY OUTCOMES:
Safety and tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Manicourt, MD, PhD, Study Director — Department of Rheumatology, University hospital St Luc, Brussels, Belgium
Locations (1):
- St Luc University Hospital, Department of Rheumatology, Université Catholique de Louvain, Brussels, Belgium